CLINICAL TRIAL: NCT06049121
Title: In Vivo Biofilm Accumulation on Implants With 3 Different Surfaces
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Andreas Stavropoulos, Professor, Malmö University
Other Study IDs: 1
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Peri-Implantitis
Keywords: Biofilm; Peri-implantitis; In vivo; Implantoplasty
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A frequent sequela of peri-implantitis itself, but also of its surgery, is the exposure of the implant surface to the oral environment. This moderately-rough surface with threads, when exposed to the oral environment, is difficult to clean. Therefore, in cases where the implant surface is expected to remain exposed or to be in direct contact with the peri-implant mucosa, implantoplasty has been proposed to obtain a smoother surface. A smoother surface should allow more efficient plaque control. This in vivo study aims to evaluate potential differences in terms of plaque accumulation between 3 different implant surfaces.

Ten participants will wear the removable splint carrying 2 implants of each type of surface (i.e., turned, modified, and modified treated with implantoplasty) for 3 days and they will be asked to remove it to perform their (usual) oral hygiene and immerse the device in cold-tap water. On day 3, the removable splint will be collected for analysis. The area of biofilm covering the implants will be quantified with different methods.

DETAILED DESCRIPTION:
The aim of this in vivo study is to evaluate potential differences in terms of plaque accumulation among 3 different implant surfaces (i.e., turned, modified, and modified treated with implantoplasty).

Splint fabrication At the first visit, a maxillary alginate impression and a gypsum cast will be produced for every participant. This cast will be used to build a removable vacuum splint, which in turn will allow to carry six implants during the study period (i.e., 2 implants of each group T, M, I). Both on the right- and left-buccal aspects of the cast, three implants (i.e., 1 implant of each group T, M, I) will be randomly allocated and secured in their position prior to making the vacuum splint. The splint will be individually trimmed and polished to provide both retention and comfort.

At the second visit, splints will be tried and, if necessary, adjusted to avoid any discomfort. Participants will be instructed in detail on how to wear and handle the splint.

At the third visit, splints will be collected and stored for analyses.

Sample size calculation The only previous study with a similar study design (Azzola et al., 2020) included only a single participant. Based on the presented data of this specific study and due to the large difference between the test and control group, a reasonable sample size calculation was not feasible. Thus, a sample size of 10 participants was arbitrarily chosen for the present study.

Ethical Considerations All splints will be individually adapted, and implants will be fixated on the buccal aspect to avoid any interference while speaking. Also, mucosal and gingival irritation will be avoided by polishing the splints on the edges and keeping a distance from the gingival margin. Further, as participants will be instructed to remove the splint to brush and floss their teeth on a regular basis, there will be no increased risk of caries or gingivitis due to biofilm accumulation during the 3-day study period.

ELIGIBILITY:
Inclusion Criteria:

* adults, > 18 years old
* systemically healthy
* full mouth healthy periodontal conditions

Exclusion Criteria

* current pregnancy or breastfeeding
* heavy smokers (> 10 cigarettes per day)
* antibiotic intake in the previous 3 months
* orthodontic appliances in the upper jaw
* removable prosthesis in the upper jaw
* extensive implant-supported restorations in the upper jaw
* active carious lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited at the Faculty of Odontology of Malmö University after informed consent is obtained
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
quantification of the biofilm | 3 days
  Quantification with crystal violet biofilm quantification assay

CONTACTS AND LOCATIONS:
Locations (1):
- Malmö University, Malmo, Sweden

REFERENCES:
- [Derived] Bertl K, Al-Said M, Mourad A, Mayol M, Lopes da Silva Z, Papia E, Stavropoulos A. Reduced Biofilm Accumulation on Implants Treated With Implantoplasty-An In Situ Trial With a Within-Subject Comparison. Clin Exp Dent Res. 2024 Dec;10(6):e70043. doi: 10.1002/cre2.70043. PMID 39610010